CLINICAL TRIAL: NCT02368223
Title: Feasibility of a Home-based Interactive System for Upper Limb Therapy (YouGrabber)
Brief Title: Feasibility of the Portable YouGrabber System
Acronym: YouGrabber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YouGrabber_Feasibility_2014
Record Dates: First submitted 2015-02-13; First posted 2015-02-23 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Cerebral Palsy; Stroke; Traumatic Brain Injury; Meningomyelocele; Central Nervous System Diseases
Keywords: Children; Rehabilitation; Telerehabilitation; Upper limb therapy
MeSH Terms: conditions — Cerebral Palsy; Stroke; Brain Injuries, Traumatic; Meningomyelocele; Central Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- YouGrabber training (Experimental): Home-based YouGrabber training
  Interventions: Device: YouGrabber

INTERVENTIONS:
Device: YouGrabber — 2 weeks of home-based therapy with a virtual-reality enhanced upper limb training system

SUMMARY:
The aim of the study is to determine the feasibility of the portable version of the YouGrabber® system in children with central motor disorders.

DETAILED DESCRIPTION:
In a feasibility trial with the portable version of the YouGrabber® system it will be determined if the technique and equipment are ready to be used in a home setting where children with central motor disorders train with assistance of caregivers but without a therapist. Furthermore, it will be examined if children and adolescents with central motor disorders accept this home-based system and if they are motivated for using it.

ELIGIBILITY:
Inclusion Criteria:

* Central motor disorders
* Ability to sit in an upright position for 45 minutes

Exclusion Criteria:

* Manual Ability Classification Scale (MACS) V
* Severe visual or auditory impairments
* Severe photosensitive epilepsy

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
User satisfaction (Questionnaire about usability, motivation, general opinion) | week 2
  Questionnaire about usability, motivation, general opinion

SECONDARY OUTCOMES:
Device usage (Total time of exercise per week; time of training session) | week 2
  Total time of exercise per week; time of training session
Error rate (Error prone games; application problems as a home-based system) | week 2
  Error prone games; application problems as a home-based system

CONTACTS AND LOCATIONS:
Overall Officials: Corinna Gerber, MSc, Principal Investigator — University Children's Hospital Zurich, Rehabilitation Centre Affoltern am Albis
Locations (1):
- University Children's Hospital Zurich, Rehabilitation Centre Affoltern am Albis, Affoltern am Albis, Switzerland

REFERENCES:
- [Derived] Gerber CN, Kunz B, van Hedel HJ. Preparing a neuropediatric upper limb exergame rehabilitation system for home-use: a feasibility study. J Neuroeng Rehabil. 2016 Mar 23;13:33. doi: 10.1186/s12984-016-0141-x. PMID 27008504